CLINICAL TRIAL: NCT01720849
Title: Efficiency of 4-aminopyridin (Fampyra) on Gait, Vision, Cognition, Fatigue and Micturation in Patients With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: FampyraCSS
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Sclerosis; EDSS 4-7
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Fampyra group
  Interventions: Drug: Fampyra

INTERVENTIONS:
Drug: Fampyra — The will be given as per normal patient treatment plan

SUMMARY:
The aim of the study is to assess improvement in visual evoked potential, cognition, fatigue, micturation and walking impairment under 3 months of Fampyra treatment

ELIGIBILITY:
Inclusion Criteria:

All patients who according to the compound's Norwegian prescription guidelines are deemed eligible for the study, i.e. MS patients with impaired walking as determined by an EDSS 4-7. They do not need a past history of optic neuritis, cognitive failure, fatigue or difficulties micturating.

Exclusion Criteria:

MS patients with contraindications to the compound according to the prescription guidelines.

Patients who have been exposed to Fampyra in the past Patients with an MS attack within last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who according to the compound's Norwegian prescription guidelines are deemed eligible for the study, i.e. MS patients with impaired walking as determined by an EDSS 4-7. They do not need a past history of optic neuritis, cognitive failure, fatigue or difficulties micturating.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
change from baseline in visual evoked potential after 2 weeks and 3 months | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vestre Viken Helseforetak, Drammen, Norway